CLINICAL TRIAL: NCT06853522
Title: A Randomized, Single-blind Clinical Study of Human Umbilical Cord Mesenchymal Stem Cell Exosomes for the Treatment of Moderate-to-severe Active Ulcerative Colitis After Existing Therapy Failure
Brief Title: hucMSCs Exosomes for the Treatment of Active Ulcerative Colitis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025YS-004
Record Dates: First submitted 2025-02-13; First posted 2025-03-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exos Localized Treatment Group (Experimental): The corresponding exosome content of 60×10^6 umbilical cord mesenchymal stem cells was given
  Interventions: Drug: exosomes derived from human umbilical cord mesenchymal stem cells
- Placebo Localized Treatment Group (Placebo Comparator): Equal amount of saline +5% albumin
  Interventions: Drug: saline +5% albumin

INTERVENTIONS:
Drug: exosomes derived from human umbilical cord mesenchymal stem cells — The corresponding exosome content of 60×10^6 umbilical cord mesenchymal stem cells was given
  Other Names: exosomes
  Arms: Exos Localized Treatment Group
Drug: saline +5% albumin — Equal amount of saline +5% albumin was given
  Other Names: placebo
  Arms: Placebo Localized Treatment Group

SUMMARY:
To evaluate the safety and efficacy of hUC-MSCs-Exos in the treatment of ulcerative colitis.

DETAILED DESCRIPTION:
A large number of previous studies and literature data collection have demonstrated the efficacy of hUC-MSCs-Exos in animal models of inflammatory bowel disease, so the investigators will further verify the safety and effectiveness of hUC-MSCs-Exos in the treatment of UC patients, and provide new ideas for clinical treatment of UC.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have had UC for at least 3 months (since symptom onset). The diagnosis should be confirmed by clinical and endoscopic evidence and confirmed by histopathological reports (note: if no previous reports are available, endoscopy and histopathology may be performed at the time of screening).
2. Subjects had active UC, defined as four-component Mayo score of 6-12 (inclusive), endoscopy score ≥2, rectal bleeding score ≥1, and bowel frequency score ≥1.
3. 18 to 75 years old, weight ≥40 kg
4. Meet at least one of the following a/b/c criteria: a. inadequate or non-response to one or more of the following treatments: i) oral prednisone ≥40mg/ day (or equivalent) or budesonide ≥9mg/ day or equivalent or beclomethasone ≥5mg/ day for at least 2 weeks. ii) At least 8 weeks of immunomodulators (AZA≥2 mg/kg/ day or 6-MP≥1.0mg/kg/ day [or lower doses, but 6-thioguanine nucleotides with therapeutic concentrations recorded]). iii) Oral administration of aminosalicylate (e.g. Mesalazine, salazine sulfopyridine, oxalazine, balsalazine) in accordance with the dosage and duration of the applicable local instructions. iv) The frontier therapy for UC has completed at least the induction dosing regimen, At doses greater than or equal to the approved instructions: anti-TNF anti-integrins (e.g., Vederizumab), JAK inhibitors (e.g., Tofaciib, Upatinib, or filgotinib), anti-IL-23 or anti-IL-12/23 drugs for the treatment of UC (e.g., ulinumab), S1PR modulators (e.g., ozamod) b. Corticosteroid dependence: failure to taper successfully to <10mg/ day of prednisone or equivalent or <6mg/ day of budesonide or <5mg/ day of beclometasone within 3 months of starting treatment (i.e., disease onset), or relapse occurs within 3 months of stopping corticosteroids. c. Intolerance to 1 or 2 of the following treatments (e.g., inability to reach the therapeutic dose or duration of treatment due to dose-limiting adverse reactions) i) corticosteroids: Adverse reactions associated with dose-limiting therapy may include, but are not limited to, infections, hyperglycemia, osteoporosis, insomnia, or psychiatric disorders. ii) Immunomodulators: Adverse reactions associated with dose-restricted therapeutic administration may include, but are not limited to, infection, nausea/vomiting, fatigue, myelosuppression, or liver toxicity.
5. Being treated with any of the following permitted drugs during the study period and meeting the drug stabilization requirements (if applicable): a. Oral corticosteroids must be stable for at least 2 weeks before randomization at an equivalent dose of ≤20 mg prednisone or ≤9mg budesonide or ≤5mg beclomethasone per day. b. A steady dose of oral aminosalicylate should be maintained for at least 2 weeks before randomization. c.AZA, 6-MP, or MTX(≤15 mg/ week) should be maintained at a stable dose for at least 4 weeks before randomization.
6. Participate voluntarily and sign a written informed consent. -

Exclusion Criteria:

1. Diagnosis of CD or undefined colitis (IBD- undefined) or other types of colitis or enteritis that may confuse assessment of effectiveness.
2. The current diagnosis is explosive colitis and/or toxic megacolon.
3. Had received fecal microbial transplantation within 4 weeks prior to randomization.
4. Had been hospitalized for UC within 2 weeks prior to screening.
5. There is clear evidence of past or current low or high grade colon dysplasia, including dysplasia detected during screening colonoscopy that has not been completely resectable.
6. Have any active or severe infection that does not resolve after adequate treatment.
7. Hepatitis B, hepatitis C virus infection, tuberculosis, HIV, uncontrollable diabetes, mental illness.
8. Have undergone organ transplantation requiring sustained immunosuppressive therapy.
9. A history of cancer within the past 5 years (except for completely treated non-melanoma skin cell carcinoma or carcinoma in situ of the cervix after complete surgical removal). Subjects who have had a diagnostic evaluation that suggests malignancy (e.g., chest or breast imaging) and who cannot reasonably rule out malignancy after additional clinical evaluation will be excluded from this study.
10. A history of drug or alcohol abuse in the 6 months prior to screening (as reported by the subject).

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2027-04-04 (Estimated); Study Completion 2028-04-04 (Estimated)

PRIMARY OUTCOMES:
Mayo Score | Baseline, 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The complete Mayo Score consists of four assessments, each scored on a scale of 0 to 3: stool frequency, rectal bleeding, endoscopy, and the physician's global assessment (PGA) of disease activity. The endoscopy subscore of the complete Mayo Score is derived from the central reading of endoscopy results by a qualified central laboratory. Patient-reported stool frequency and rectal bleeding, as well as the PGA reported by the clinician, will be collected in an electronic diary.

SECONDARY OUTCOMES:
Geboes Score | Baseline, at 12 weeks after treatment.
  It is the most commonly used histological scoring system for colonic mucosa in the field of ulcerative colitis (UC). It is divided into six grades: 1) Structural changes (Grade 0); 2) Chronic inflammatory infiltration (Grade 1); 3) Neutrophils and eosinophils in the lamina propria (Grade 2); 4) Neutrophils in the epithelium (Grade 3); 5) Crypt destruction (Grade 4); 6) Erosion or ulceration (Grade 5). Each grade is further divided into four subcategories. The Geboes score ranges from 0 to 5.4, with higher scores indicating more severe inflammation. Typically, active histological inflammation in UC is defined as a Geboes score of ≥2B.1.
Inflammatory Bowel Disease Questionnaire (IBDQ) | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The IBDQ is a well-established assessment tool for measuring disease-specific health-related quality of life. It consists of 32 items : bowel symptoms (10 items), systemic symptoms (5 items), emotional functioning (12 items), and social functioning (5 items). The questionnaire is scored using a 7-point Likert scale, ranging from worst health (1) to best health (7). Domain scores are calculated by summing the item responses, with higher values indicating better quality of life.The total score range of the IBDQ is 32-224, which can be obtained by adding up the scores of individual domains. According to the total score, a meaningful change in the IBDQ score (also defined as an IBDQ response) is defined as a change of ≥ 16 points, and this threshold has been applied in studies involving subjects with Crohn's disease (CD) or ulcerative colitis (UC). In addition, IBDQ remission can be defined as a total score of ≥ 170 points.
The item of urgency to defecate | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  Subjects are required to complete a single item that assesses how frequently they needed to empty their bowels immediately to avoid an accident in the past 7 days. The response scale ranges from 0 (never) to 4 (more than once a day).
EQ-5D-5L | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The EQ-5D-5L is a brief self-report measure of health status and function. The descriptive system of this instrument includes 5 items for measuring problems (none, mild, moderate, severe, or extreme), covering mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In total, the responses to these items describe 5^5 = 3,125 health states. The responses of the subjects to the 5 items can be weighted and aggregated to generate a utility index score that measures the social value of their current health. These scores range from 1 (perfect health) to 0 (death), and negative values indicate a health state worse than death. Additionally, the EQ-5D-5L includes a Visual Analogue Scale (VAS), which allows subjects to rate their current health on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
  Among patients receiving treatment for IBD, a meaningful change in the EQ-5D-5L VAS score is defined as a change of ≥ 10 points.
CRP (C - reactive protein) | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The unit for CRP is milligrams per liter (mg/L), with the normal reference value typically being ≤10 mg/L.When there is a bacterial infection, the CRP level usually increases significantly, which can exceed 100 mg/L, or even be higher. In contrast, when there is a viral infection, the CRP level generally does not increase or only increases slightly, usually not exceeding 50 mg/L. Therefore, CRP testing can be used to distinguish between bacterial infections and viral infections. The CRP level is positively correlated with the severity of the infection. The more severe the infection is, the more obvious the increase in CRP will be. By monitoring the changes in the CRP level, the therapeutic effect of the infection treatment and the progression of the disease can be evaluated.
fecal calprotectin | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The unit for fecal calprotectin is micrograms per gram of stool (μg/g), with a normal range of 0-50 μg/g. Values exceeding this range may indicate intestinal inflammation or disease activity (such as in inflammatory bowel disease).
immune cell subsets | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The detection of immune cell subsets (such as T cells, B cells, and NK cells) is usually expressed as a percentage (%).
BMI (Body Mass Index) | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The unit is kilograms per square meter (kg/m²). It is calculated using the formula: weight (kg) ÷ height² (m²). Normal range: 18.5-24 kg/m² (for adults).
albumin | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The unit is grams per liter (g/L). It reflects liver synthetic function and nutritional status. Normal reference values are 35-50 g/L for adults and 34-48 g/L for individuals aged 60 years or older.
Hemoglobin | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The unit is grams per liter (g/L). It is used to assess anemia or polycythemia. Normal reference values are as follows: adult males: 120-160 g/L; adult females: 110-150 g/L.
body temperature | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The unit is degrees Celsius (℃). Normal range: axillary temperature is 36℃ to 37℃.
Respiratory Rate | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The unit is breaths per minute (breaths/min). Normal range: adults, 16-20 breaths/min (at rest).Tachypnea may be caused by reasons such as pneumonia, fever, cardiovascular diseases, anemia, etc., while bradypnea may be caused by reasons such as increased intracranial pressure, hypothyroidism, etc.
Blood Pressure | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The unit is millimeters of mercury (mmHg). Normal range: systolic pressure, 90-139 mmHg; diastolic pressure, 60-89 mmHg.
Heart Rate | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The unit is beats per minute (beats/min). Normal range: 60-100 beats/min (at rest).
Blood White Blood Cells | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  Normal range for adults is 4.0-10.0×10⁹/L. An elevated level may indicate bacterial infection or inflammation, while a decreased level may be associated with viral infections or drug reactions.
Bloos Red Blood Cells | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  Normal range is 4.3-5.8×10¹²/L for males and 3.8-5.1×10¹²/L for females.
Platelets | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  Normal range is 125-350×10⁹/L. A reduced count increases the risk of bleeding, while an elevated count increases the risk of thrombosis.
Urine White Blood Cells | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  The reference value of white blood cells is 0 to 5 cells per high-power field (HP). If the number of white blood cells in each high-power field exceeds 5, it is called pyuria under the microscope, which suggests the possible presence of infections or other pathological changes in the urinary system.
Urine Red Blood Cells | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  Under normal circumstances, the number of urinary red blood cells is 0-3 per high-power field (HP). If the number of urinary red blood cells in each high-power field exceeds 3, it is called microscopic hematuria.
Urinary Protein | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  Normal value is negative (-).The test results of urinary protein are affected by various factors. For example, strenuous exercise, fever, a high-protein diet, etc., may all lead to a transient increase in physiological urinary protein, which can return to normal after removing the influencing factors. It may also indicate the presence of kidney diseases and other conditions.
occult blood test (OB) | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  Normally, the result is negative. A positive result is commonly seen in hemorrhagic diseases of the digestive tract.
alanine aminotransferase (ALT) | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  Normal range is 7-40 U/L. Elevated levels indicate liver damage.
aspartate aminotransferase (AST) | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  Normal range is 13-35 U/L. Elevated levels indicate liver damage.
serum creatinine (Cr) | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  Normal range is 53-106 μmol/L for males and 44-97 μmol/L for females. Elevated levels suggest decreased renal function.
Blood Urea Nitrogen (BUN) | Baseline, at 1 week, 4 weeks, 8 weeks, and 12 weeks after treatment.
  Normal range is 2.9-7.5 mmol/L. Elevated levels may be associated with renal failure or dehydration.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No